CLINICAL TRIAL: NCT05649943
Title: APPROACH : Multimodal Approach in Patients With mHSPC. A Pragmatic Randomized Trial of Apalutamide Plus Androgen Deprivation Therapy (APA-ADT) Versus APA-ADT Plus Local Treatment. A Meet-URO 29 Study
Brief Title: Multimodal Approach in Patients With mHSPC. Randomized Trial of APA+ADT vs APA-ADT and Local Treatment
Acronym: APPROACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: ASST Santi Paolo e Carlo (Other); European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
MeSH Terms: interventions — Glutamyl Aminopeptidase; Androgen Antagonists; apalutamide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA + ADT + RP/RT (Other): Apalutamide 240 mg, four 60 mg tablets as an oral single daily dose, according to clinical practice, plus Androgen Deprivation Therapy (ADT) plus clinician-driven choice local treatment with Radiotherapy or Radical Prostatectomy, six months after starting treatment with apalutamide
  Interventions: Drug: APA + ADT; Procedure: Local Treatmetn RT or RP
- APA + ADT (Other): Apalutamide 240 mg, four 60 mg tablets as an oral single daily dose, according to clinical practice, plus Androgen Deprivation Therapy (ADT)
  Interventions: Drug: APA + ADT

INTERVENTIONS:
Drug: APA + ADT — All participants will receive apalutamide 240 mg (4 x 60 mg) tablets orally once daily. Apalutamide is distributed in Italy under the trade name of Erleada® 60 mg.
  All patients not undergoing surgical castration should also continue medical castration by taking a gonadotropin-releasing hormone (GnRHa) analogue during treatment.
  Other Names: Apalutamide 240 mg + Androgen Deprivation Therapy
Procedure: Local Treatmetn RT or RP — Patients who will undergo radiotherapy as a local treatment must be treated according to the following scheme:
  External beam radiotherapy administered at 36 Gy in six consecutive weekly fractions of 6 Gy, or 55 Gy in 20 daily fractions of 2・75 Gy over 4 weeks.
  Radiation therapy will be given with the patient supine and with a full bladder and an empty rectum. The planned target volume is prostate only, with an 8 mm margin posteriorly and a 10 mm margin elsewhere.
  No RT on lymph nodes is foreseen. RT should begin 6 months after the first dose of apalutamide (+/- 2 weeks).
  Radical prostatectomy should be performed 6 months after the first dose of apalutamide (+/- 2 weeks).
  Other Names: Local treatment with radiotherapy or radical prostatectomy, clinician-driven choice
  Arms: APA + ADT + RP/RT

SUMMARY:
Italian multicenter study, will enroll ~566 pts with oligometastatic hormone sensitive prostate cancer who are candidates to receive treatment with apalutamide.

After 6 months from the start of treatment, patients will be randomized to receive local treatment based on the investigator's choice ( either one between primary radiotherapy or cytoreductive prostatectomy), in addition to apalutamide, or to continue just with medical therapy.

DETAILED DESCRIPTION:
Primary end point: To determine whether treatment with apalutamide in combination with androgen-deprivative therapy for 6 months followed by locoregional treatment with radiotherapy or radical prostatectomy has better efficacy than medical treatment with apalutamide + ADT alone in terms of radiographic progression-free survival (rPFS), specifically time to radiographic progression in soft tissue per RECIST 1.1 or in bone per PCWG3 criteria by investigator, or death. Secondary end points: To evaluate tumor shrinkage after locoregional approach and to evaluate short and long term side effects after locoregional surgery or RT, time to PSA progression, time to castration resistance, cancer specific survival, overall survival and quality of life according to EPIC-26 and EQ-5D-5L questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically confirmed diagnosis of prostate adenocarcinoma
* Metastatic disease documented by ≥1 bone lesion with Technetium 99m (99mTc) bone scan. Individuals with only one bone lesion should have confirmation of that lesion on CT or MRI.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) Grade ≤ 2
* No previous treatment with antiandrogens or GnRH analogues, or a treatment ≤ 3 months.
* No previous systemic or local treatment for prostate adenocarcinoma, including pelvic radiotherapy.
* Laboratory values at the time of screening:

  a. Neutrophils ≥ 1500/μL b. Hemoglobin ≥ 9.0 mg/μL (no transfusions in the past 28 days) c. Platelets ≥ 100,000/μL d. Creatinine ≤ 2 x upper limit of normal and serum albumin ≥ 3.0 g/dL f. Total bilirubin ≤ 1.5 x upper limit of normal [NOTE: In subjects with Gilbert syndrome, if total bilirubin is >1.5 x ULN, measure direct and indirect bilirubin, and if direct bilirubin is ≤ 1.5 x ULN subjects may be eligible]; g. AST and ALT ≤ 2.5 x upper limit of normal
* Able to swallow Apalutamide tablets whole.
* All subjects must sign an Informed Consent Form indicating that they understand the purpose of the study and its procedures and intend to participate. The subject must be willing and must be able to comply with the restrictions specified in this protocol.

Inclusion criteria for cytoreductive surgery:

* Age >18 years
* Clinical stage cT3
* Robot-assisted radical prostatectomy with iliac obturator lymphadenectomy
* Surgical piece management criteria similar to Proteus criteria.

Exclusion Criteria:

* Pathologic findings consistent with small cell, ductal, or neuroendocrine prostate cancer.
* Known brain metastases.
* Lymph node metastases only.
* Visceral metastases.
* Patients not eligible for surgery or radiotherapy.
* Unacceptable increase in cardiovascular risk, defined as the occurrence of at least one of the following episodes in the 6 months prior to randomization: unstable angina, myocardial infarction, symptomatic congestive heart failure, clinically significant thromboembolic events (e.g., pulmonary embolism), or clinically significant ventricular arrhythmias .
* Uncontrolled high blood pressure (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg).
* Previous treatment with antiandrogens, GnRH analogues, or other systemic treatments for adenocarcinoma of the prostate.
* Previous local treatment with surgery and/or radiotherapy.
* Any prior malignancy (except adequately treated basal cell carcinoma or a squamous cell skin carcinoma, superficial bladder carcinoma, or any other in situ carcinoma currently in complete remission) within 5 years of randomization.
* Known allergies, hypersensitivity or intolerance to the excipients of Apalutamide.
* Patients who, within 28 days prior to randomisation, have received:

  1. transfusions (red blood cells and/or platelets);
  2. hematopoietic growth factors;
  3. major surgery.
* Symptomatic and/or chronic viral hepatitis; chronic liver disease; moderate or severe liver failure (class B and C according to the Child-Pugh scale); encephalopathy, ascites or thrombo-haemorrhagic disorders secondary to liver failure.
* Gastrointestinal disorders affecting drug absorption
* Active infections requiring systemic therapy such as human immunodeficiency virus (HIV);
* Any condition or situation which, in the judgment of the investigator, precludes participation in this trial.

Exclusion criteria for cytoreductive surgery:

* Contraindication for surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) | Up to 48 months
  Evaluation of the efficacy of treatment with APA+ADT for 6 months followed by locoregional treatment with radiotherapy or radical prostatectomy compared to treatment with APA+ ADT alone in terms of Radiographic Progression-Free Survival (rPFS) in patients with hormone prostate adenocarcinoma -susceptible with low-volume metastatic disease.

SECONDARY OUTCOMES:
Local event - free survival | Up to 48 months
  Defined as the absence of one of the following conditions in the follow up: urinary retention, hydronephrosis, acute or chronic renal failure exacerbation, intestinal obstruction
Local treatment - free survival | Up to 48 months
  Defined as the absence of the need for one of the following interventions: trans-urethral resection of the prostate, placement of a ureteral stent or nephrostomy for hydronephrosis, bladder catheterization, surgery for intestinal obstruction/colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Guadalupi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (3):
- Italy (3):
  - European Institute of Oncology, Milan, Lombardy
  - ASST Santi Paolo e Carlo, Milan, Lombardy
  - Istituto Tumori Milano, Milan, Mi

REFERENCES:
- [Background] Chi KN, Agarwal N, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez Soto A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Deprince K, Naini V, Li J, Cheng S, Yu MK, Zhang K, Larsen JS, McCarthy S, Chowdhury S; TITAN Investigators. Apalutamide for Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2019 Jul 4;381(1):13-24. doi: 10.1056/NEJMoa1903307. Epub 2019 May 31. PMID 31150574
- [Background] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, De Porre P, Smith AA, Brookman-May SD, Li S, Zhang K, Rooney B, Lopez-Gitlitz A, Small EJ. Apalutamide and Overall Survival in Prostate Cancer. Eur Urol. 2021 Jan;79(1):150-158. doi: 10.1016/j.eururo.2020.08.011. Epub 2020 Sep 6. PMID 32907777
- [Background] Metcalfe MJ, Smaldone MC, Lin DW, Aparicio AM, Chapin BF. Role of radical prostatectomy in metastatic prostate cancer: A review. Urol Oncol. 2017 Apr;35(4):125-134. doi: 10.1016/j.urolonc.2017.01.001. Epub 2017 Feb 9. PMID 28190749
- [Background] Mathieu R, Korn SM, Bensalah K, Kramer G, Shariat SF. Cytoreductive radical prostatectomy in metastatic prostate cancer: Does it really make sense? World J Urol. 2017 Apr;35(4):567-577. doi: 10.1007/s00345-016-1906-3. Epub 2016 Aug 8. PMID 27502935
- [Background] Gravis G, Boher JM, Joly F, Soulie M, Albiges L, Priou F, Latorzeff I, Delva R, Krakowski I, Laguerre B, Rolland F, Theodore C, Deplanque G, Ferrero JM, Culine S, Mourey L, Beuzeboc P, Habibian M, Oudard S, Fizazi K; GETUG. Androgen Deprivation Therapy (ADT) Plus Docetaxel Versus ADT Alone in Metastatic Non castrate Prostate Cancer: Impact of Metastatic Burden and Long-term Survival Analysis of the Randomized Phase 3 GETUG-AFU15 Trial. Eur Urol. 2016 Aug;70(2):256-62. doi: 10.1016/j.eururo.2015.11.005. Epub 2015 Nov 21. PMID 26610858
- [Background] Inaba K, Tsuchida K, Kashihara T, Umezawa R, Takahashi K, Okuma K, Murakami N, Ito Y, Igaki H, Sumi M, Nakayama Y, Shinoda Y, Hara T, Matsui Y, Komiyama M, Fujimoto H, Itami J. Treatment results of radiotherapy to both the prostate and metastatic sites in patients with bone metastatic prostate cancer. J Radiat Res. 2021 May 12;62(3):511-516. doi: 10.1093/jrr/rraa056. PMID 33822986
- [Background] Heidenreich A, Pfister D, Porres D. Cytoreductive radical prostatectomy in patients with prostate cancer and low volume skeletal metastases: results of a feasibility and case-control study. J Urol. 2015 Mar;193(3):832-8. doi: 10.1016/j.juro.2014.09.089. Epub 2014 Sep 22. PMID 25254935
- [Background] Culp SH, Schellhammer PF, Williams MB. Might men diagnosed with metastatic prostate cancer benefit from definitive treatment of the primary tumor? A SEER-based study. Eur Urol. 2014 Jun;65(6):1058-66. doi: 10.1016/j.eururo.2013.11.012. Epub 2013 Nov 20. PMID 24290503
- [Background] Sooriakumaran P, Karnes J, Stief C, Copsey B, Montorsi F, Hammerer P, Beyer B, Moschini M, Gratzke C, Steuber T, Suardi N, Briganti A, Manka L, Nyberg T, Dutton SJ, Wiklund P, Graefen M. A Multi-institutional Analysis of Perioperative Outcomes in 106 Men Who Underwent Radical Prostatectomy for Distant Metastatic Prostate Cancer at Presentation. Eur Urol. 2016 May;69(5):788-94. doi: 10.1016/j.eururo.2015.05.023. Epub 2015 May 30. PMID 26038098
- [Background] Gratzke C, Engel J, Stief CG. Role of radical prostatectomy in metastatic prostate cancer: data from the Munich Cancer Registry. Eur Urol. 2014 Sep;66(3):602-3. doi: 10.1016/j.eururo.2014.04.009. Epub 2014 May 10. No abstract available. PMID 24821581
- [Background] Leyh-Bannurah SR, Gazdovich S, Budaus L, Zaffuto E, Briganti A, Abdollah F, Montorsi F, Schiffmann J, Menon M, Shariat SF, Fisch M, Chun F, Steuber T, Huland H, Graefen M, Karakiewicz PI. Local Therapy Improves Survival in Metastatic Prostate Cancer. Eur Urol. 2017 Jul;72(1):118-124. doi: 10.1016/j.eururo.2017.03.020. Epub 2017 Apr 3. PMID 28385454
- [Background] Heidenreich A, Fossati N, Pfister D, Suardi N, Montorsi F, Shariat S, Grubmuller B, Gandaglia G, Briganti A, Karnes RJ. Cytoreductive Radical Prostatectomy in Men with Prostate Cancer and Skeletal Metastases. Eur Urol Oncol. 2018 May;1(1):46-53. doi: 10.1016/j.euo.2018.03.002. Epub 2018 May 15. PMID 31100228
- [Background] Parker CC, James ND, Brawley CD, Clarke NW, Hoyle AP, Ali A, Ritchie AWS, Attard G, Chowdhury S, Cross W, Dearnaley DP, Gillessen S, Gilson C, Jones RJ, Langley RE, Malik ZI, Mason MD, Matheson D, Millman R, Russell JM, Thalmann GN, Amos CL, Alonzi R, Bahl A, Birtle A, Din O, Douis H, Eswar C, Gale J, Gannon MR, Jonnada S, Khaksar S, Lester JF, O'Sullivan JM, Parikh OA, Pedley ID, Pudney DM, Sheehan DJ, Srihari NN, Tran ATH, Parmar MKB, Sydes MR; Systemic Therapy for Advanced or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Radiotherapy to the primary tumour for newly diagnosed, metastatic prostate cancer (STAMPEDE): a randomised controlled phase 3 trial. Lancet. 2018 Dec 1;392(10162):2353-2366. doi: 10.1016/S0140-6736(18)32486-3. Epub 2018 Oct 21. PMID 30355464
- [Background] Van den Broeck T, Oprea-Lager D, Moris L, Kailavasan M, Briers E, Cornford P, De Santis M, Gandaglia G, Gillessen Sommer S, Grummet JP, Grivas N, Lam TBL, Lardas M, Liew M, Mason M, O'Hanlon S, Pecanka J, Ploussard G, Rouviere O, Schoots IG, Tilki D, van den Bergh RCN, van der Poel H, Wiegel T, Willemse PP, Yuan CY, Mottet N. A Systematic Review of the Impact of Surgeon and Hospital Caseload Volume on Oncological and Nononcological Outcomes After Radical Prostatectomy for Nonmetastatic Prostate Cancer. Eur Urol. 2021 Nov;80(5):531-545. doi: 10.1016/j.eururo.2021.04.028. Epub 2021 May 5. PMID 33962808